CLINICAL TRIAL: NCT07355842
Title: Role of Slow Waves in the Progression of Neurodegeneration in Isolated REM Sleep Behavior Disorder
Acronym: SloW-iRBD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: University Hospital, Zürich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SloW-iRBD; 2025-D0069 (Other: BASEC)
Record Dates: First submitted 2025-12-22; First posted 2026-01-21 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Parkinson Disease; REM Sleep Behavior Disorder (iRBD)
Keywords: Parkinson; Parkinson disease; Sleep; Neurodegeneration; Auditory stimulation; iRBD; REM sleep behavior disorder
MeSH Terms: conditions — Parkinson Disease; REM Sleep Behavior Disorder; Nerve Degeneration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum arm (Experimental): Nightly enhancement of slow waves through Phase Targeted Auditory Stimulation (PTAS) over 18 months.
  Interventions: Device: Tosoo Axora
- Sham arm (Sham Comparator): Nightly application of tones that will be applied in a non-PTAS manner, resulting in no enhancement of slow waves over 18 months.
  Interventions: Device: Tosoo Axora

INTERVENTIONS:
Device: Tosoo Axora — Phase Targeted Auditory Stimulation (PTAS) will be applied through integrated headphones with a portable EEG device when non-rapid-eye-movement (NREM) sleep is detected during the night.
  Other Names: PTAS Intervention (Verum)
  Arms: Verum arm
Device: Tosoo Axora — Auditory stimuli will be delivered during the night through integrated headphones with a portable EEG device in a non-PTAS manner.
  Other Names: PTAS Intervention (Sham)
  Arms: Sham arm

SUMMARY:
This study tests whether enhancing deep sleep with gentle sounds at night can slow progression in people with iRBD or early Parkinson's disease. Participants wear a sensor headband and headphones for 18 months. Four assessments including mobility, memory, imaging (PET/MRI), lumbar puncture, and blood tests are assessed.

DETAILED DESCRIPTION:
Many people with REM sleep behavior disorder (iRBD) develop Parkinson's disease or similar conditions over the years. To date, there is no effective method to prevent this transition. Animal experiments and observational studies in patients and older adults indicate that deeper sleep is associated with a slower progression of brain changes. In this study, we are now investigating whether enhancement of deep sleep using sounds during sleep can influence the progressive brain changes in iRBD or early Parkinson's disease.

Participants wear a headband with sensors and headphones for 18 months, which plays gentle sounds during sleep to enhance deep sleep. In addition, four examinations are carried out, including tests of mobility, memory, imaging (PET/MRI), a lumbar puncture, and blood sampling. Two of the examinations will take place at the University Hospital of Zurich, and two more can also be carried out at home if desired.

The aim is to investigate whether enhancement of deep sleep can help slow the progression of iRBD or early-stage Parkinson's disease. The study is double-blind and controlled, which means that neither the participants nor the researchers know who is receiving the active treatment.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Diagnosis of polysomnography-confirmed isolated REM Sleep Behavior Disorder (iRBD) based on international criteria (ICSD-3), combined with EITHER
* UPDRS III without action tremor ≥ 4 AND abnormal olfaction, OR
* diagnosis of PD along international criteria for less than 2 years

Further inclusion criteria are:

* no dopaminergic treatment and no foreseen start of such treatment during duration of the study
* ability to apply the intervention, alone or with help of a co-habitant, stable living situation
* sufficient language skills in German, French or Italian
* negative pregnancy test for women of child-bearing potential

Exclusion Criteria:

* Suspected or known non-compliance to other therapies
* current or recent participation in another clinical trial
* extended absences
* hearing impairment that prevents hearing the tones for auditory stimulation
* non-responder to auditory stimulation during screening
* clinically significant concomitant disease or unstable condition
* Apnea-Hypopnea-Index (AHI) > 15/h or under Continuous Positive Airway Pressure (CPAP) treatment
* Restless Legs Syndrome
* meeting criteria for diagnosis of atypical Parkinson syndrome
* diagnosis of Dementia or Montreal Cognitive Assessment (MoCA) < 24
* severe Depression or other psychiatric disorder
* regular use of benzodiazepines and other central nervous system depressant substances
* current or recent history within the last year of substance abuse disorders or chronic alcohol consumption
* recent or planned major surgery
* history of allergies and hypersensitivity relevant for electrode application or medication allergies
* additional exclusion criteria for PET imaging
* any criterion that may pose the participant at risk
* breastfeeding, intention to become pregnant, or unwillingness to use medically reliable contraception for women of child-bearing potential

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Presynaptic Dopaminergic Integrity | assessed at Baseline Visit and Closeout Visit (after 18 months)
  Striatal dopaminergic function as measured by high-resolution 18F-Fluorodopa (18F-DOPA)-PET imaging.

SECONDARY OUTCOMES:
MDS-UPDRS Part III Score | assessed at each visit (Baseline, after 6 months, after 12 months, after 18 months (Closeout))
  Motor symptom severity assessed by the Movement Disorder Society-Unified Parkinson's Disease Rating Scale Part III (MDS-UPDRS III), a clinician-rated examination of motor signs.
Purdue Pegboard Test Score | assessed at each visit (Baseline, after 6 months, after 12 months, after 18 months (Closeout))
  Manual dexterity and fine motor coordination assessed by total score on the Purdue Pegboard Test.
Alternate Finger Tapping Test | assessed at each visit (Baseline, after 6 months, after 12 months, after 18 months (Closeout))
  Motor speed and coordination assessed by performance on the Alternate Finger Tapping Test.
UPDRS I.1 (subjective cognition) | assessed at each visit (Baseline, after 6 months, after 12 months, after 18 months (Closeout))
  Patient-reported cognitive experiences of daily living assessed by MDS-UPDRS Part I, Item 1.1.
Montreal Cognitive Assessment (MoCA) Score | assessed at each visit (Baseline, after 6 months, after 12 months, after 18 months (Closeout)
  Global cognitive function assessed by MoCA total score.
Trail Making Test Part A | assessed at each visit (Baseline, after 6 months, after 12 months, after 18 months (Closeout))
  Processing speed and attention assessed by time to completion on Trail Making Test Part A.
Trail Making Test Part B | assessed at each visit (Baseline, after 6 months, after 12 months, after 18 months (Closeout))
  Executive function assessed by time to completion on Trail Making Test Part B.
Digit Span Forward | assessed at each visit (Baseline, after 6 months, after 12 months, after 18 months (Closeout))
  Attention assessed by Digit Span Forward from the Wechsler Adult Intelligence Scale.
Digit Span backward | assessed at each visit (Baseline, after 6 months, after 12 months, after 18 months (Closeout))
  Working memory assessed by Digit Span Backward from the Wechsler Adult Intelligence Scale
Stroop Test | assessed at each visit (Baseline, after 6 months, after 12 months, after 18 months (Closeout))
  Executive function and inhibitory control assessed by Stroop Color-Word Test.
Verbal Fluency - Semantic | assessed at each visit (Baseline, after 6 months, after 12 months, after 18 months (Closeout))
  Semantic verbal fluency assessed by category fluency task.
Benton Judgment of Line Orientation (BJLO) | assessed at each visit (Baseline, after 6 months, after 12 months, after 18 months (Closeout))
  Visuospatial function assessed by Benton Judgment of Line Orientation test.
LPS-4 Logical Reasoning | assessed at Baseline Visit and Closeout Visit (after 18 months)
  Logical reasoning assessed by Leistungsprüfsystem subtest 4.
Rey-Taylor Complex Figure Test - Copy | assessed at Baseline Visit and Closeout Visit (after 18 months)
  Visuoconstruction assessed by copy trial of the Rey-Taylor Complex Figure Test.
Rey-Taylor Complex Figure Test - Recall | assessed at Baseline Visit and Closeout Visit (after 18 months)
  Visual memory assessed by delayed recall of the Rey-Taylor Complex Figure Test.
California Verbal Learning Test (CVLT) | assessed at Baseline Visit and Closeout Visit (after 18 months)
  Verbal learning and memory assessed by California Verbal Learning Test.
Verbal Fluency - Phonemic | assessed at Baseline Visit and Closeout Visit (after 18 months)
  Phonemic verbal fluency assessed by letter fluency task.
Boston Naming Test (BNT) | assessed at Baseline Visit and Closeout Visit (after 18 months)
  Naming and language function assessed by Boston Naming Test
WAIS Similarities | assessed at Baseline Visit and Closeout Visit (after 18 months)
  Verbal abstract reasoning assessed by similarities subtest from the Wechsler Adult Intelligence Scale

OTHER OUTCOMES:
Exploratory Outcome: Home Sleep EEG - Sleep Microstructure | Continuous over 18 months
  NREM sleep oscillatory activity and microstructural features measured by portable EEG device (Tosoo Axora) during nightly use, including but not limited to slow wave activity, sleep spindles, and their temporal dynamics.
Exploratory Outcome: Home Sleep EEG - Sleep Macrostructure | Continuous over 18 months
  Sleep architecture and derived metrics measured by portable EEG device (Tosoo Axora) during nightly use, including sleep stage distribution, sleep continuity, and sleep timing parameters.
Exploratory Outcome: MRI | assessed at Baseline Visit and Closeout Visit (after 18 months)
  Neuroanatomical and vascular markers assessed by brain MRI, including structural imaging, phase-contrast imaging, arterial spin labeling, and related sequence
Exploratory Outcome: 18F-DOPA PET - Exploratory Parameters | assessed at Baseline Visit and Closeout Visit (after 18 months)
  Exploratory PET parameters including visual assessment of striatal uptake patterns, influx constant (Ki), and F-DOPA distribution beyond predefined regions of interest
Exploratory Outcome: Psychomotor Vigilance Task (PVT) | assessed at each visit (Baseline, after 6 months, after 12 months, after 18 months (Closeout))
  Sustained attention and reaction time assessed by the Psychomotor Vigilance Task.
Exploratory Outcome: Sustained Attention to Response Task (SART) | assessed at each visit (Baseline, after 6 months, after 12 months, after 18 months (Closeout))
  Vigilance and response inhibition assessed by the Sustained Attention to Response Task.
Exploratory Outcome: Glucose Metabolism | assessed at Baseline Visit and Closeout Visit (after 18 months)
  Glucose metabolism (HbA1c, glycosylated hemoglobin) will be assessed to explore glucose tolerance and control through a simple blood draw.
Exploratory Outcome - Polysomnography - Sleep Architecture | assessed at Baseline Visit and Closeout Visit (after 18 months)
  Sleep macrostructure including total sleep time, sleep efficiency, and sleep stage distribution assessed by in-laboratory polysomnography.
Exploratory Outcome: Polysomnography - REM Sleep Without Atonia | assessed at Baseline and Closeout (18 months)
  REM sleep without atonia (RWA) quantified as percentage of REM sleep with elevated muscle tone on polysomnography.
Exploratory Outcome: Actigraphy - Sleep-Wake Patterns | assessed before/after each visit (Baseline, after 6 months, after 12 months, Closeout (18 months)) for 2 weeks each
  Sleep-wake rhythm including total sleep time, sleep efficiency, and rest-activity patterns assessed by wrist actigraphy over 2-week periods.
Exploratory Outcome: Sleep Diary | Assessed before/after each visit (Baseline, after 6 months, after 12 months, Closeout (18 months)) for 2 weeks each
  Self-reported sleep timing, duration, and quality recorded daily over 2-week periods.
Exploratory Outcome: Sleep Quality- Visual Analog Scale - | assessed before/after each visit (Baseline, after 6 months, after 12 months, Closeout (18 months)) for 2 weeks each
  Subjective sleep quality assessed by Visual Analog Scale.
Exploratory Outcome - Karolinska Sleepiness Scale (KSS) | assessed before/after each visit (Baseline, after 6 months, after 12 months, Closeout (18 months)) for 2 weeks each
  Subjective daytime sleepiness assessed by Karolinska Sleepiness Scale.
Exploratory Outcome: Retinal Nerve Fiber Layer Thickness (RNFL) | assessed at Baseline Visit and Closeout Visit (after 18 months)
  Retinal nerve fiber layer thickness measured by optical coherence tomography (OCT)
Exploratory Outcome: Ganglion Cell-Inner Plexiform Layer Thickness (GCIPL) | assessed at Baseline Visit and Closeout Visit (after 18 months)
  Ganglion cell-inner plexiform layer thickness measured by optical coherence tomography (OCT)
Exploratory Outcome: Macular Vessel Density (MVD) | assessed at Baseline Visit and Closeout Visit (after 18 months)
  Macular vessel density measured by optical coherence tomography angiography (OCT-A)
Exploratory Outcome: Non-Motor Symptoms Scale (NMSS) | assessed at each visit (Baseline, after 6 months, after 12 months, after 18 months (Closeout))
  Non-motor symptom severity and frequency assessed by the Non-Motor Symptoms Scale, a 30-item questionnaire covering nine symptom dimensions
Exploratory Outcome: Epworth Sleepiness Scale (ESS) | assessed at each visit (Baseline, after 6 months, after 12 months, after 18 months (Closeout))
  Daytime sleepiness assessed by the Epworth Sleepiness Scale (8-item self-report questionnaire)
Exploratory Outcome: Parkinson's Disease Sleep Scale-2 (PDSS-2) | assessed at each visit (Baseline, after 6 months, after 12 months, after 18 months (Closeout))
  Sleep disturbances assessed by the PDSS-2, a 15-item self-administered questionnaire covering motor problems at night, PD-specific nocturnal symptoms, and disturbed sleep.
Exploratory Outcome: Ikelos Rating Scale | assessed at each visit (Baseline, after 6 months, after 12 months, after 18 months (Closeout))
  RBD symptom severity assessed by the Ikelos Rating Scale, evaluating frequency and severity of REM sleep behavior disorder
Exploratory Outcome: Exploratory Outcome: EQ-5D-5L | assessed at each visit (Baseline, after 6 months, after 12 months, after 18 months (Closeout))
  Health-related quality of life assessed by the EQ-5D-5L questionnaire, covering mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, plus visual analogue scale
Exploratory Outcome: Blood Biomarkers | assessed at Baseline Visit and Closeout Visit (after 18 months)
  Neurodegenerative and inflammatory markers measured in blood, including neurofilament light chain (NfL) and alpha-synuclein
Exploratory Outcome: CSF Biomarkers | assessed at Baseline Visit and Closeout Visit (after 18 months)
  Neurodegenerative and inflammatory markers measured in cerebrospinal fluid, including amyloid-β, tau, alpha-synuclein, and neurofilament light chain (optional, for participants who consent to lumbar puncture)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Luft, Prof. Dr. med., Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Neurology Department, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No